CLINICAL TRIAL: NCT05153785
Title: Intravenous Lidocaine for Postoperative Recovery in Liver Surgery, a Randomized Double Blinded Placebo-controlled Study
Brief Title: Perioperative Intravenous Lidocaine in Liver Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lidokain vid leverkirurgi; 2019-002361-35 (EudraCT Number)
Record Dates: First submitted 2021-11-12; First posted 2021-12-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Liver Metastases; Liver Cancer; Postoperative Pain; Opioid Use
Keywords: liver surgery; postoperative pain; Lidocaine; opioid use
MeSH Terms: conditions — Liver Neoplasms; Pain, Postoperative | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized double blinded placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine arm (Experimental): The experimental arm will receive a bolus of 1,5mg/kg Lidocaine before induction of anesthesia, immediately followed by an infusion of 1,5mg/kg/h until 1 hour post surgery.
  Interventions: Drug: Lidocaine
- Placebo arm (Placebo Comparator): The placebo arm will receive the same amount of normal Saline.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — Intravenous perioperative Lidocain for pain Control and improvement of postoperative recovery
  Arms: Lidocaine arm
Drug: Normal saline — Placebo
  Arms: Placebo arm

SUMMARY:
This is a randomized double blinded placebo-controlled study, conducted in Lund, Sweden. Patients will be randomized in two groups, with a ratio of 1:1. The experimental arm will receive intravenous Lidocaine perioperatively, and the Control arm will receive placebo, i.e. normal Saline. Postoperative both arms will get routine pain Control with PCA, Patient Controlled Analgesia with an intravenous Oxycodone-infusion. Outcome-measures will include patients pain intensity scoring, and opioid consumption.

DETAILED DESCRIPTION:
Patientes will be randozied in blocks of eight.

The experimental arm will receive a bolus of 1,5mg/kg before induction of anesthesia, immediately followed by an infusion of 1,5mg/kg/h until 1 hour post surgery. The placebo arm will receive the same amount of normal Saline instead. Pain intensity scoring, measured by Numerical Rating Scale, NRS, will be conducted at 1, 2, 4 hour postoperatively, and each morning and night until discharge, or for a maximum 5 Days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 yy
* Patient planned for minor hepatectomy
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Cirrosis
* ASA>3
* Elevated liver enzymes
* AV-block >1, without pacemaker
* WHO class >2
* Allergy against Lidocain or other amid-type local anasthesia
* Heart failure
* Epilepsy
* Treatment with class III anti-arythimic medication
* Preoperative ongoing opioid usage
* Use of : Erythromycin, clarithromycin, Fluvoxamine, Cimetidine, ciprofloxacin, antivirala-HIV-läkemedel or imidazol the week before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Opioid consumption at 24 hours | 24 hours postoperatively
  Sum of opioids consumed

SECONDARY OUTCOMES:
Opioid consumption at 48 hours | 48 hours postoperatively
  Sum of opioids consumed
Opioid consumption at 72 hours | 72 hours postoperatively
  Sum of opioids consumed
Opioid consumption at 96 hours | 96 hours postoperatively
  Sum of opioids consumed
Opioid consumption at 120 hours | 120 hours postoperatively
  Sum of opioids consumed
Postoperative pain intensity | Day 0-5 postoperatively, twice every day
  Numerical rating scale (NRS) in rest and activity, scale 0-10, 0=no pain, 10=worst imaginable pain
Number of participants with Postoperative comlications | 30 days postoperatively
  Comparition of Complications classified according to Clavien Dindo, 0,1,2,3a,3b,4,5
Level of Postoperative comlications | 30 days postoperatively
  Complications classified according to Clavien Dindo, 0,1,2,3a,3b,4a,4b,5, 0 beeing none and 5 beeng death.
Time to return of Bowel function | Day 0-30 postoperatively
  Time to first flatus and defacation
Number of participants with Postoperative nausea and vomiting | Day 1-5 postopertively
  Postoperative nausea and vomiting, as noted in questionary "Quality of recovery-40"
Level of Postoperative nausea and vomiting | Day 1-5 postopertively
  Postoperative nausea and vomiting, as noted in questionary "Quality of recovery-40"
Days in hospital | 0-90 days postoperatively
  Length of hospital stay
Level of MEGX concentrations | Twice during surgery, and once 1 hour after surgery.
  Concentration of the metabolite "MEGX" in patients blood
Level of Lidocaine concentration | Twice during surgery, and once 1 hour after surgery.
  Concentration of Lidocaine in patients blood
Mortality | 30 days postoperatively
  death after surgery
Rating of Quality of recovery-40 | Day 1-5 postoperatively
  Quality of recovery questionary.
Number of participant with Adverse Events | 0-30 days
  All adverse events
Level of adverse events | 0-30 days
  All adverse events, classified according to CTCEA
Number of participants with Chronic Postsurgical pain | 3 months after surgery
  Chronic Postsurgical pain, according to Brief Pain inventory- questionary
Level of Chronic Postsurgical pain | 3 months after surgery
  Chronic Postsurgical pain, according to Brief Pain inventory- questionary

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Tingstedt, Prof, Study Director — Lund University Hospital
Locations (1):
- Skåne University Hospital of Lund, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication, for 10 years.

REFERENCES:
- [Background] Sun Y, Li T, Wang N, Yun Y, Gan TJ. Perioperative systemic lidocaine for postoperative analgesia and recovery after abdominal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2012 Nov;55(11):1183-94. doi: 10.1097/DCR.0b013e318259bcd8. PMID 23044681
- [Background] Marret E, Rolin M, Beaussier M, Bonnet F. Meta-analysis of intravenous lidocaine and postoperative recovery after abdominal surgery. Br J Surg. 2008 Nov;95(11):1331-8. doi: 10.1002/bjs.6375. PMID 18844267
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Background] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Background] Weibel S, Jelting Y, Pace NL, Helf A, Eberhart LH, Hahnenkamp K, Hollmann MW, Poepping DM, Schnabel A, Kranke P. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery in adults. Cochrane Database Syst Rev. 2018 Jun 4;6(6):CD009642. doi: 10.1002/14651858.CD009642.pub3. PMID 29864216
- [Background] Kranke P, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Weibel S. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. Cochrane Database Syst Rev. 2015 Jul 16;(7):CD009642. doi: 10.1002/14651858.CD009642.pub2. PMID 26184397
- [Background] Dunn LK, Durieux ME. Perioperative Use of Intravenous Lidocaine. Anesthesiology. 2017 Apr;126(4):729-737. doi: 10.1097/ALN.0000000000001527. No abstract available. PMID 28114177
- [Background] Yardeni IZ, Beilin B, Mayburd E, Levinson Y, Bessler H. The effect of perioperative intravenous lidocaine on postoperative pain and immune function. Anesth Analg. 2009 Nov;109(5):1464-9. doi: 10.1213/ANE.0b013e3181bab1bd. PMID 19843784
- [Background] Ortiz MP, Godoy MC, Schlosser RS, Ortiz RP, Godoy JP, Santiago ES, Rigo FK, Beck V, Duarte T, Duarte MM, Menezes MS. Effect of endovenous lidocaine on analgesia and serum cytokines: double-blinded and randomized trial. J Clin Anesth. 2016 Dec;35:70-77. doi: 10.1016/j.jclinane.2016.07.021. Epub 2016 Aug 6. PMID 27871598
- [Background] Sridhar P, Sistla SC, Ali SM, Karthikeyan VS, Badhe AS, Ananthanarayanan PH. Effect of intravenous lignocaine on perioperative stress response and post-surgical ileus in elective open abdominal surgeries: a double-blind randomized controlled trial. ANZ J Surg. 2015 Jun;85(6):425-9. doi: 10.1111/ans.12783. Epub 2014 Jul 31. PMID 25078385
- [Background] Kuo CP, Jao SW, Chen KM, Wong CS, Yeh CC, Sheen MJ, Wu CT. Comparison of the effects of thoracic epidural analgesia and i.v. infusion with lidocaine on cytokine response, postoperative pain and bowel function in patients undergoing colonic surgery. Br J Anaesth. 2006 Nov;97(5):640-6. doi: 10.1093/bja/ael217. Epub 2006 Sep 4. PMID 16952918
- [Background] Moore PA, Hersh EV. Local anesthetics: pharmacology and toxicity. Dent Clin North Am. 2010 Oct;54(4):587-99. doi: 10.1016/j.cden.2010.06.015. PMID 20831923
- [Background] Rosenberg PH, Veering BT, Urmey WF. Maximum recommended doses of local anesthetics: a multifactorial concept. Reg Anesth Pain Med. 2004 Nov-Dec;29(6):564-75; discussion 524. doi: 10.1016/j.rapm.2004.08.003. PMID 15635516
- [Background] Cassuto J, Wallin G, Hogstrom S, Faxen A, Rimback G. Inhibition of postoperative pain by continuous low-dose intravenous infusion of lidocaine. Anesth Analg. 1985 Oct;64(10):971-4. PMID 3898920
- [Background] Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, Hering W. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesth Analg. 2004 Apr;98(4):1050-1055. doi: 10.1213/01.ANE.0000104582.71710.EE. PMID 15041597
- [Background] Herroeder S, Pecher S, Schonherr ME, Kaulitz G, Hahnenkamp K, Friess H, Bottiger BW, Bauer H, Dijkgraaf MG, Durieux ME, Hollmann MW. Systemic lidocaine shortens length of hospital stay after colorectal surgery: a double-blinded, randomized, placebo-controlled trial. Ann Surg. 2007 Aug;246(2):192-200. doi: 10.1097/SLA.0b013e31805dac11. PMID 17667496
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Martin F, Cherif K, Gentili ME, Enel D, Abe E, Alvarez JC, Mazoit JX, Chauvin M, Bouhassira D, Fletcher D. Lack of impact of intravenous lidocaine on analgesia, functional recovery, and nociceptive pain threshold after total hip arthroplasty. Anesthesiology. 2008 Jul;109(1):118-23. doi: 10.1097/ALN.0b013e31817b5a9b. PMID 18580181
- [Background] Striebel HW, Klettke U. [Is intravenous lidocaine infusion suitable for postoperative pain management?]. Schmerz. 1992 Dec;6(4):245-50. doi: 10.1007/BF02527813. German. PMID 18415635
- [Background] Usubiaga JE, Wikinski J, Ferrero R, Usubiaga LE, Wikinski R. Local anesthetic-induced convulsions in man--an electroencephalographic study. Anesth Analg. 1966 Sep-Oct;45(5):611-20. No abstract available. PMID 5950380
- [Background] Drayer DE, Lorenzo B, Werns S, Reidenberg MM. Plasma levels, protein binding, and elimination data of lidocaine and active metabolites in cardiac patients of various ages. Clin Pharmacol Ther. 1983 Jul;34(1):14-22. doi: 10.1038/clpt.1983.122. PMID 6861434
- [Background] DeToledo JC. Lidocaine and seizures. Ther Drug Monit. 2000 Jun;22(3):320-2. doi: 10.1097/00007691-200006000-00014. PMID 10850400
- [Background] Beaussier M, Delbos A, Maurice-Szamburski A, Ecoffey C, Mercadal L. Perioperative Use of Intravenous Lidocaine. Drugs. 2018 Aug;78(12):1229-1246. doi: 10.1007/s40265-018-0955-x. PMID 30117019
- [Background] Rimback G, Cassuto J, Tollesson PO. Treatment of postoperative paralytic ileus by intravenous lidocaine infusion. Anesth Analg. 1990 Apr;70(4):414-9. PMID 2316883
- [Background] Wallin G, Cassuto J, Hogstrom S, Linden I, Faxen A, Rimback G, Hedner T. Effects of lidocaine infusion on the sympathetic response to abdominal surgery. Anesth Analg. 1987 Oct;66(10):1008-13. PMID 3631561
- [Background] De Oliveira GS Jr, Duncan K, Fitzgerald P, Nader A, Gould RW, McCarthy RJ. Systemic lidocaine to improve quality of recovery after laparoscopic bariatric surgery: a randomized double-blinded placebo-controlled trial. Obes Surg. 2014 Feb;24(2):212-8. doi: 10.1007/s11695-013-1077-x. PMID 24036842
- [Background] Dale GJ, Phillips S, Falk GL. The analgesic efficacy of intravenous lidocaine infusion after laparoscopic fundoplication: a prospective, randomized, double-blind, placebo-controlled trial. Local Reg Anesth. 2016 Dec 2;9:87-93. doi: 10.2147/LRA.S119483. eCollection 2016. PMID 27980437
- [Background] Baral BK, Bhattarai BK, Rahman TR, Singh SN, Regmi R. Perioperative intravenous lidocaine infusion on postoperative pain relief in patients undergoing upper abdominal surgery. Nepal Med Coll J. 2010 Dec;12(4):215-20. PMID 21744761
- [Background] Yon JH, Choi GJ, Kang H, Park JM, Yang HS. Intraoperative systemic lidocaine for pre-emptive analgesics in subtotal gastrectomy: a prospective, randomized, double-blind, placebo-controlled study. Can J Surg. 2014 Jun;57(3):175-82. doi: 10.1503/cjs.009613. PMID 24869609